CLINICAL TRIAL: NCT05367154
Title: Identification of Factors Related to Unintended Initial Dissection of the Posterior Plane in Small Incision Lenticule Extraction Cases by Three Different Surgeons
Brief Title: Factor Analysis of Unintended Initial Dissection of the Posterior Plane
Status: Completed | Type: Observational
Sponsor: Yifeng Yu (Other)
Responsible Party: Sponsor-Investigator, Yifeng Yu, Deputy chief physician of Ophthalmology center of the Second Affiliated Hospital of Nanchang University, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Other Study IDs: [2021] No. (031)
Record Dates: First submitted 2022-04-29; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Myopia; Small-incision Lenticule Extraction (SMILE) Surgery
Keywords: femtosecond laser; small-incision lenticule extraction (SMILE); unintended initial dissection of the posterior plane
MeSH Terms: conditions — Myopia; Smiling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eyes with SMILE surgeries: Eyes with SMILE surgeries which were performed by three surgeons with different experiences.
  Interventions: Procedure: Small incision lenticule extraction

INTERVENTIONS:
Procedure: Small incision lenticule extraction — Small incision lenticule extraction surgeries performed by two Refractive surgery experts (Refractive surgery expert 1: YYF, Associate Professor with 10 years of experience as a refractive surgeon; Refractive surgery expert 2: GF, Associate Professor with 5 years of experience as a refractive surgeon) and a Attending ophthalmologist (WNY, Attending ophthalmologist with 1 year of experience as a refractive surgeon).

SUMMARY:
To explore the potential factors for unintended initial dissection of the posterior plane in a large sample retrospective analysis and surgeons of different levels.

DETAILED DESCRIPTION:
Myopia is the most common eye disease in the world. Femtosecond laser small incision lens extraction (SMILE) has increasingly become the first choice in refractive surgery due to its greater biomechanical stability, less impact on the tear film and other advantages. However, because SMILE surgery is more challenging than flap-based corneal ablative surgery, young surgeons sometimes dissect the lenticule posterior plane first in clinical practice, which will make it more difficult to extract the lenticule or even cause the retained lenticule. The purpose of this study aims to explore the potential risk factors for unintended initial dissection of the posterior plane in large samples and surgeons of different surgical volumes and different surgical habits (different angles of peripheral corneal incision) in multiple scenarios.

ELIGIBILITY:
Inclusion Criteria:

* A condition in which the spherical equivalent refractive error of an eye is ≤ -0.50 D when ocular accommodation is relaxed;
* Age ≥18 years;
* Spherical equivalent (SE) ≥ -10.0D;
* Corrected distance visual acuity (CDVA) ≥ 16/20;
* Stable myopia for at least 2 years;
* No contact lenses wearing for at least 2 weeks.

Exclusion Criteria:

* The presence or history of eye conditions other than myopia and astigmatism, such as keratoconus or external eye injury;
* A history of eye surgery;
* The presence or history of systemic diseases.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients from clinics in ophthalmic center of the second Affiliated Hospital of Nanchang University
Sampling Method: Non-Probability Sample
Enrollment: 3003 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
The number of patients with unintended initial dissection of the posterior plane in the SMILE surgeries | Day 0
  The number of patients with unintended initial dissection of the posterior plane were observed during the SMILE surgeries.

SECONDARY OUTCOMES:
The impact of spherical equivalent on the unintended initial dissection of the posterior plane (UIDPP) in SMILE surgeries | Day 0
  The spherical equivalent of eyes with UIDPP and eyes without UIDPP were analyzed, and statistical analysis was observed to investigate the impact of spherical equivalent on the UIDPP in SMILE surgeries.
The impact of peripheral corneal incision angle on the unintended initial dissection of the posterior plane (UIDPP) in SMILE surgeries | Day 0
  The peripheral corneal incision angle of eyes with UIDPP and eyes without UIDPP were analyzed, and statistical analysis was observed to investigate the impact of peripheral corneal incision angle on the UIDPP in SMILE surgeries.
The impact of peripheral lens thickness on the unintended initial dissection | Day 0
  The peripheral lens thickness of eyes with UIDPP and eyes without UIDPP were analyzed, and statistical analysis was observed to investigate the impact of peripheral corneal incision angle on the UIDPP in SMILE surgeries.
The impact of lens diameter on the unintended initial dissection | Day 0
  The lens diameter of eyes with UIDPP and eyes without UIDPP were analyzed, and statistical analysis was observed to investigate the impact of lens diameter on the UIDPP in SMILE surgeries.
The impact of central corneal thickness on the unintended initial dissection | Day 0
  The central corneal thickness of eyes with UIDPP and eyes without UIDPP were analyzed, and statistical analysis was observed to investigate the impact of central corneal thickness on the UIDPP in SMILE surgeries.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No